CLINICAL TRIAL: NCT06184009
Title: Treatment of Newly Diagnosed High Risk Pediatric Acute Lymphoblastic Leukemia-prospective, Nationwide, Multi-center Study
Brief Title: Treatment of Newly Diagnosed High Risk Pediatric Acute Lymphoblastic Leukemia
Acronym: HR ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jae Wook Lee (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Pusan National University Yangsan Hospital (Other); Korea University Anam Hospital (Other)
Responsible Party: Sponsor-Investigator, Jae Wook Lee, Principal Investigator, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-3626-0001
Record Dates: First submitted 2023-12-05; First posted 2023-12-28 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Acute Lymphoblastic Leukemia
Keywords: HR ALL; NGS-MRD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALL, High risk with DI #2(Doxorubicin) (Experimental): * Clinical and genetic factors consistent with High risk : Induction → Consolidation
    1. BM MRD < 0.01% after both Induction and Consolidation : IM #1 → DI #1 → IM #2 → Maintenance
    2. BM MRD ≥ 0.01% after Induction, < 0.01% after Consolidation : IM #1 → DI #1 → IM #2 → DI #2 → Maintenance
    3. BM MRD ≥ 0.01% after Consolidation
    <!-- -->
    1. T cell ALL : Change to very high risk regimen
    2. Pre-B ALL : IM #1 → Intensification
       1. BM MRD < 0.01% after IM #1 : Continue with 'No. 2' of High risk regimen starting with DI #1
       2. BM MRD ≥ 0.01% after IM #1 : Change to Very high risk regimen
          * T cell ALL patients with M1 BM post-Consolidation will start IM #1. However, the patients will switch to Very high risk regimen at the next chemotherapy cycle once post-Consolidation MRD ≥ 0.01% has been reported.
  Interventions: Drug: ALL, High risk

INTERVENTIONS:
Drug: ALL, High risk — Intervention Description :
  * Clinical and genetic factors consistent with High risk : Induction → Consolidation
    1. BM MRD < 0.01% after both Induction and Consolidation : IM #1 → DI #1 → IM #2 → Maintenance
    2. BM MRD ≥ 0.01% after Induction, < 0.01% after Consolidation : IM #1 → DI #1 → IM #2 → DI #2 → Maintenance
    3. BM MRD ≥ 0.01% after Consolidation
    <!-- -->
    1. T cell ALL : Change to very high risk regimen
    2. Pre-B ALL : IM #1 → Intensification
       1. BM MRD < 0.01% after IM #1 : Continue with 'No. 2' of High risk regimen starting with DI #1
       2. BM MRD ≥ 0.01% after IM #1 : Change to Very high risk regimen
          * T cell ALL patients with M1 BM post-Consolidation will start IM #1. However, the patients will switch to Very high risk regimen at the next chemotherapy cycle once post-Consolidation MRD ≥ 0.01% has been reported.

SUMMARY:
* Clinical and genetic factors consistent with High risk : Induction → Consolidation

  1. BM MRD < 0.01% : IM #1 → DI #1 → IM #2 → Maintenance
  2. BM MRD ≥ 0.01% : IM #1 → DI #1 → IM #2 → DI #2 → Maintenance
  3. BM MRD ≥ 0.01% after Consolidation

  <!-- -->

  1. T cell ALL : Change to very high risk regimen
  2. Pre-B ALL : IM #1 → Intensification

     1. BM MRD < 0.01% after IM #1 : DI #1 → IM #2 → DI #2 → Maintenance
     2. BM MRD ≥ 0.01% after IM #1 : Change to Very high risk regimen

        * Difference in the number of 'interim maintenance(IM)' and 'delayed intensification(DI)' is important for chemotherapies based on MRD.

DETAILED DESCRIPTION:
* Clinical and genetic factors consistent with High risk : Induction → Consolidation

  1. BM MRD < 0.01% after both Induction and Consolidation : IM #1 → DI #1 → IM #2 → Maintenance
  2. BM MRD ≥ 0.01% after Induction, < 0.01% after Consolidation : IM #1 → DI #1 → IM #2 → DI #2 → Maintenance
  3. BM MRD ≥ 0.01% after Consolidation

  <!-- -->

  1. T cell ALL : Change to very high risk regimen
  2. Pre-B ALL : IM #1 → Intensification

     1. BM MRD < 0.01% after IM #1 : DI #1 → IM #2 → DI #2 → Maintenance
     2. BM MRD ≥ 0.01% after IM #1 : Change to Very high risk regimen

        * T cell ALL patients with M1 BM post-Consolidation will start IM #1. However, the patients will switch to Very high risk regimen at the next chemotherapy cycle once post-Consolidation MRD ≥ 0.01% has been reported.

ELIGIBILITY:
<Inclusion Criteria>

* Age: 1year~19years of age at diagnosis
* Patients who are newly diagnosed Pre-B ALL and meet one of the following criteria

  * High-risk group according to the National Cancer Institute (NCI)/Rome: Age greater than or equal to 10 years and less than 19 years at diagnosis, or white blood cell count greater than or equal to 50 x 10^9/L at diagnosis
  * If extra-bone marrow lesions are identified at the time of diagnosis, Central nervous system involvement (CNS3) or testicular involvement
  * High-risk gene variants:

KMT2A rearrangement intrachromosomal amplification of chromosome 21 (iAMP21)

● If subjects are under the age of 10 at the time of diagnosis and took steroids for more than 24 hours within two weeks before the diagnosis, the risk group will be determined by the presence of a whole blood test within three days before starting steroids. If a whole blood test is performed within three days before beginning steroids, the risk group will be assessed based on the white blood cell count in the test. If there is no whole blood test before starting steroids, subjects are classified as a high-risk group. If subjects are ten or older at diagnosis, pre-diagnosis steroid treatment will not affect the risk classification.

* Newly diagnosed T cell ALL

<Exclusion Criteria>

* Patients with Burkitt leukemia/lymphoma or mature B-cell leukemia
* Patients with Down syndrome
* potential of pregnancy or during pregnancy (patients of childbearing age need adequate contraception for the duration of the trial)
* Patients who have already received steroid treatment for newly diagnosed ALL specified in the above selection criteria or chemotherapies more than one intrathecal cytarabine treatment
* Participating in an interventional clinical trial other than this research

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | Up to 5 years
  Event-free survival rate for 5 years from the date of registration

SECONDARY OUTCOMES:
Overall Survival | Up to 5 years
  The time until defined by date of all-cause mortality from the date of 1st infusion
Recurred rate | Up to 5 years
  As the period from enrollment to disease progression/recurrence
Death rate related to infusion | Up to 5 years
  The time until defined by date of drug-related mortality from the date of 1st infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jae Wook Lee, Ph.D, Study Chair — The Catholic University of Korea
Locations (7):
- South Korea (7):
  - Seoul National University Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul saint Mary's Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No